CLINICAL TRIAL: NCT03128177
Title: Mechanisms of Nocturnal Hypertension and Non-Dipping Blood Pressure Patterns
Brief Title: Nocturnal Hypertension and Non-Dipping Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, David Calhoun, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F150508004
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: nocturnal hypertension; non-dipping blood pressure; obstructive sleep apnea
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Sodium, Dietary

STUDY DESIGN:
Intervention Model Description: Crossover study of high (6 g) and low (1.5 g) sodium diet
Who Masked: Participant, Investigator
Masking Description: Both the participant and investigator are blinded to the diet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High sodium diet (Experimental): High sodium diet is 6 g sodium per day for 10 days
  Interventions: Dietary Supplement: Dietary sodium
- Low sodium diet (Experimental): Low sodium diet is 1.5 g sodium per day for 10 days
  Interventions: Dietary Supplement: Dietary sodium

INTERVENTIONS:
Dietary Supplement: Dietary sodium — High (6 g) versus low (1.5 g) sodium diet

SUMMARY:
The purpose of this study is to determine if high salt diet contributes to high nighttime blood pressure. The investigators will determine if high compared to low salt diet increases 24-hour blood pressure levels. The investigators will also determine if high salt diet affects blood vessel stiffness, cardiac output, and sleep apnea. The study will also determine how high salt diet affects the activity of certain genes related to control of blood pressure. A total of 60 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Nocturnal hypertension

Exclusion Criteria:

* Stage 2 clinic hypertension
* History of congestive heart failure
* Chronic kidney disease,
* Diabetes with insulin use
* History of a cardiovascular event
* Pregnant or nursing
* Current use of continuous positive airway pressure
* Shift work
* A known circadian rhythm disorder

Ages: 48 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
24-hour blood pressure | Baseline to 7 days after start of dietary period
  Blood pressure measured by an ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Obstructive sleep apnea | Baseline to 7 days after start of dietary period
  Severity of obstructive sleep apnea as determine by the apnea hypopnea index

CONTACTS AND LOCATIONS:
Overall Officials: David Calhoun, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- David A. Calhoun, MD, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No